CLINICAL TRIAL: NCT03827460
Title: Sex Differences in the Response to Abstinence From Alcohol.
Acronym: SPAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Martin Plawecki, Assistant Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1809467722; R01AA027236-05 (NIH)
Record Dates: First submitted 2018-11-12; First posted 2019-02-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Alcoholism; Sex Differences; Abstinence; Alcohol Deprivation Effect
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Arms 1 and 2: 2 session parallel, random order, no blind.
  Arm 3: Sequential, includes all subjects who complete Arm1 or Arm 2
Masking Description: The intervention is 2 weeks of monitored abstinence from alcohol compared to usual drinking. Thus, it is not possible to mask conditions for participants or investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Free access alcohol self-administration (Experimental): During the 2.5-hour free-access self-administration sessions, the participant may choose to complete a task for an alcohol or water reward. Interventions include Abstinence from Alcohol and Usual Drinking
  Interventions: Behavioral: Abstinence from alcohol; Behavioral: Usual drinking; Drug: Intravenous Alcohol
- Clamped alcohol exposure (Experimental): A battery of behavioral tasks will be administered to participants before, and at the beginning and end of a 3 hour clamped exposure to alcohol (fixed at 80 mg/dL). EEG will be recorded throughout to assess event related potentials associated with task performance. Interventions include Abstinence from Alcohol and Usual Drinking.
  Interventions: Behavioral: Abstinence from alcohol; Behavioral: Usual drinking; Drug: Intravenous Alcohol
- 2 year followup (No Intervention): Participants from both Arm 1 and Arm 2 will be surveyed every 2 months for alcohol consumption for 2 years following the Experimental phase. Interventions include Abstinence from Alcohol and Usual Drinking.

INTERVENTIONS:
Behavioral: Abstinence from alcohol — Participants will undergo a laboratory alcohol infusion session that terminates 2 weeks of monitored abstinence from alcohol
  Arms: Clamped alcohol exposure; Free access alcohol self-administration
Behavioral: Usual drinking — Participants will undergo a laboratory alcohol infusion session during a period of usual drinking behavior
  Arms: Clamped alcohol exposure; Free access alcohol self-administration
Drug: Intravenous Alcohol — During the laboratory alcohol infusion sessions, alcohol is infused through an indwelling catheter.
  Other Names: 6.0& (v/V) ethanol solution
  Arms: Clamped alcohol exposure; Free access alcohol self-administration

SUMMARY:
In laboratory animals, repeated cycles of abstinence from and return to alcohol drinking can lead to changes in alcohol intake. In a study of the effect of abstinence on drinking in humans, the investigators found evidence that abstinence affects drinking differently in women compared to men. In the present study, the investigators propose to study how men and women respond to abstinence, and whether this information can be used to improve intervention and prevention strategies.

DETAILED DESCRIPTION:
Women and men differ in how quickly they progress from social to problematic alcohol drinking. In laboratory animals, short-term abstinence increases alcohol consumption, with repeated deprivations leading to disordered drinking. In a preliminary study, the investigators found that men and women differed in how their motivation to drink alcohol changed after a short period of abstinence. The investigators hypothesize that this difference may affect their transition to alcohol use disorders. The objectives of this application are to characterize the human post abstinence response, and use identical alcohol exposures to study the mechanisms underlying identified sex differences. In addition, the investigators will complete a 2 year prospective study of natural drinking patterns to assess how self-reported abstinence intervals influence drinking trajectories. The long-term goal of this project is to inform alcohol use disorder treatment and to design and test novel interventions using the laboratory model of post-abstinence response. There is a critical unfilled need to understand sex differences in disease progression, and this lab-based assessment coupled to longitudinal follow-up provides the rigorous experimental design to begin to meet that need. This project will increase scientific knowledge by advancing the translation between preclinical and clinical models, eventually informing sex-specific intervention and prevention strategies for problematic drinking and establishing a model to test those interventions..

ELIGIBILITY:
Inclusion Criteria:

* Moderate social drinkers
* Able to understand/complete questionnaires and procedures in English
* Body mass index (BMI) between 18.5 and 32 kg/m2
* Have venous access sufficient to allow blood sampling

Exclusion Criteria:

* Pregnant or breast-feeding women, or women who intend to become pregnant
* Do not attest to using accepted forms of birth control for the infusion phase of the study
* Current treatment for, or desire to be treated for, any substance use disorder or court ordered to not drink alcohol
* History of significant adverse reaction to alcohol
* Medical disorders or other conditions such as alcohol withdrawal seizures or delirium tremens that may influence study outcome or participant safety
* Medications (past 30 days) that could influence data or participant safety (e.g. antidepressants, antipsychotics, benzodiazepines, etc.) as determined by investigators
* DSM 5 Disorders (non AUD) or current/history of neurological disease of cerebral origin, or head injury with > 20 min loss of consciousness
* Positive breath alcohol reading on arrival at any study visit
* Actively suicidal (for example, any suicide attempts within the past year or any current suicidal intent, including a plan) or are at serious suicidal risk, by clinical judgment of the investigator
* Any condition for which the principal investigators determine it is unsafe or not prudent to enroll

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Sex differences in the effect of abstinence on alcohol self-administration. | 2 single day laboratory sessions, one following 2 weeks alcohol abstinence
  The effect of 2 weeks abstinence on intravenous alcohol intake will be compared in men and women.
Sex differences in the effect of abstinence on sensitivity of the P3 response to alcohol. | 2 single day laboratory sessions, one following 2 weeks alcohol abstinence
  The effect of 2 weeks abstinence from alcohol on sensitivity of the neurophysiological P3 response to alcohol, assessed using a stop-signal response task, will be compared in women and men during an iv infusion clamp.
Sex differences in the effect of abstinence on subjective responses to alcohol. | 2 single day laboratory sessions, one following 2 weeks alcohol abstinence
  The effect of 2 weeks abstinence from alcohol on subjective responses to alcohol in women and men will be assessed using a survey during an iv infusion clamp.
The role of changes in alcohol elimination on sex differences in response to abstinence. | 2 single day laboratory sessions, one following 2 weeks alcohol abstinence
  The effect of 2 weeks abstinence from alcohol on alcohol elimination in men and women will be assessed using an iv alcohol infusion clamp.
Response to abstinence as a predictor of alcohol risk in women and men. | 2 years
  For both Arm 1 and Arm 2, daily alcohol consumption will be surveyed every 2 months for 2 years following the laboratory sessions. Self-imposed periods of abstinence will be assessed to determine if subsequent daily alcohol intake increases or decreases, and to determine if men and women differ in the effect of abstinence on drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Plawecki, MD, PhD, Principal Investigator — Psychiatry, Indiana University School of Medicine; Melissa A Cyders, PhD, Principal Investigator — Psychology, Indiana University-Purdue University at Indianapolis
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The final raw dataset will be available to other researchers when we have collected all subjects and completed our own planned analyses. Prior to completion of our own planned analyses, we would be willing to consider releasing the dataset upon request. We will work with our IRB to establish a strategy for de-identifying the data while retaining the ability to ensure the quality of the stored data, and develop a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After all subjects have been collected and the primary outcomes accepted for publication. The dataset will be available indefinitely,
Access Criteria: On request to the PIs